CLINICAL TRIAL: NCT02652234
Title: A Single-arm, Open-label Study to Investigate the Safety, Tolerability and Pharmacokinetics of Endostar Subcutaneous Injection in Chinese Advanced NSCLC Patients
Brief Title: Study of Endostar Subcutaneous Injection in NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-ED-201504
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: NSCLC
MeSH Terms: interventions — endostar protein; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endostar-subcutaneous injection/Chemotherapy (Experimental)
  Interventions: Drug: Endostar; Drug: Chemotherapy

INTERVENTIONS:
Drug: Endostar — Endostar, ih, QD，day 1 of cycle 1; Endostar, ih, QD，day 2-15 of cycle 3;
Drug: Chemotherapy

SUMMARY:
This is an open-label, single-arm study to assess the safety, tolerability and pharmacokinetics of Endostar subcutaneous injection in Chinese advanced NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological confirmed unresectable stage ⅢB～Ⅳ non-squamous NSCLC
* ECOG performance status 0-1
* Life expectancy≥3 months
* Adequate hematologic function: WBC≥3.0×109/L ,ANC≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L;
* Adequate hepatic and renal function: ALT≤2.5×ULN, AST≤2.5×ULN, TBIL≤1.5×ULN, creatinine≤1×ULN, creatinine clearance≥50ml/min;
* Normal coagulation function (PT, APTT, TT, Fbg) ;
* Patients signed informed consent form;
* Willingness and capability to comply with protocol requirement and well communicate with investigators.

Exclusion Criteria:

* With uncontrolled ascites or pleural effusion;
* Patients receiving a chest or abdominal surgery within 28 days before enrollment; or with not fully healed surgical incision; or expected to receive surgery during the study;
* History of ischemic or TIA within 6 months before enrollment;
* Uncontrolled hypertension, hypertensive crisis or hypertensive encephalopathy;
* Arrhythmias need to be treated; history of coronary artery disease (including angina pectoris and myocardial infarction) or ischemic myocardium; congestive heart-failure NYHA class ≥ II；
* Serious active infections;
* History of abdominal fistula, gastrointestinal perforation, abdominal abscess within 6 months prior to enrollment;
* Symptomatic brain or meningeal metastasis;
* Epileptic seizure need to be treated;
* HCV, HBV or HIV positive;
* History of other malignant tumors within 5 years (except curable cervix carcinoma in situ or skin basal cell carcinoma);
* Known allergies to any excipient in the study drug;
* Any conditions that may interfere with the patient's participation in the study or have an impact on the assessment of the results of the study;
* Any conditions that may endanger patient safety or interfere with the patient's compliance;
* Pregnant and lactating women;
* The investigators consider the patients unsuitable for this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
incidence of adverse events | until 30 days after the last dose

SECONDARY OUTCOMES:
Cmax | day1, day2 of cycle1;day1,day2,day4,day13,day14,day15,day16,day17 of cycle2; day2,day13,day14,day15 of cycle3; up to 9 weeks
AUC | day1, day2 of cycle1;day1,day2,day4,day13,day14,day15,day16,day17 of cycle2; day2,day13,day14,day15 of cycle3; up to 9 weeks
Tmax | day1, day2 of cycle1;day1,day2,day4,day13,day14,day15,day16,day17 of cycle2; day2,day13,day14,day15 of cycle3; up to 9 weeks
T1/2 | day1, day2 of cycle1;day1,day2,day4,day13,day14,day15,day16,day17 of cycle2; day2,day13,day14,day15 of cycle3; up to 9 weeks
CL | day1, day2 of cycle1;day1,day2,day4,day13,day14,day15,day16,day17 of cycle2; day2,day13,day14,day15 of cycle3; up to 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jia Chen, MD, Principal Investigator — Jiangsu Province Cancer Hospital; Lingxiang Chen, MD, Principal Investigator — Jiangsu Province Cancer Hospital
Locations (1):
- Jiangsu Province Cancer Hospital, Nanjing, Jiangsu, China